CLINICAL TRIAL: NCT00975546
Title: Intrauterine Insemination for HIV-discordant Couples
Brief Title: HIV-discordant Couple Intrauterine Insemination
Status: No longer available | Type: Expanded Access
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Erma Drobnis, Clinical Asssistant Professor, University of Missouri-Columbia
Other Study IDs: HIV-IUI
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Infertility; HIV Infections
Keywords: fertility; HIV discordant; HIV; Infertility in HIV-discordant couples; HIV seronegativity
MeSH Terms: conditions — Infertility; HIV Infections

INTERVENTIONS:
Other: Sperm washing and testing for HIV contamination — Semen will undergo specialized washing to reduce viral contamination of sperm. The sperm are first separated from leukocytes and other seminal constituents by centrifugation over a stepwise gradient. Motile sperm will be separated from the resulting pellet by a swim-up step in which washed sperm are overlaid with fresh medium into which sperm migrate. The final sperm suspension will be stored while testing for HIV is performed by reverse transcription polymerase chain reaction (RT-PCR)
Procedure: Intrauterine Insemination — Intrauterine Insemination (IUI) will be performed on the HIV-negative wife, following standard clinical practice, using washed sperm from her HIV-positive husband after testing the IUI sample for HIV.

SUMMARY:
The investigators propose to treat couples who wish to have a child in which the man is HIV-positive and the woman is HIV-negative. The investigators call these couples HIV-discordant. On the average, an HIV-positive man, who does not participate in high-risk activities, will transmit HIV to a female partner one in every one thousand acts of intercourse without a condom. To reduce transmission of HIV, HIV-discordant couples are counseled to avoid intercourse altogether, or to use condoms during every act of intercourse. In order to have a child, these patients can use donor insemination. If they wish to have a natural child of the infected man, they can use a combination of medication of the man to reduce the amount of virus in his semen, and condom use except at the time of ovulation when the woman produces an egg. This reduces the chance of infecting the woman, but studies have shown that about 4% of women will be infected with HIV using this approach. Alternatively, they can use vitro fertilization (IVF) with intra cytoplasmic sperm injection (ICSI) in which eggs are collected from the woman after hormone-stimulation and are fertilized in the laboratory by injecting a single washed sperm from her husband into each egg. The resulting embryos can be transferred to the wife's uterus and/or frozen for later use. These procedures are believed to minimize the risk of HIV transmission (although the number of cases is low), but IVF-ICSI is very expensive and are not an option for everyone. A simpler method used for over 15 years in Europe is to collect the man's semen, wash the sperm in the laboratory, and test the sperm sample for HIV before placing it in the woman's uterus (intrauterine insemination; IUI). Although the risk of HIV transmission to the woman is presumably not zero with this method, over 4000 inseminations reported have not resulted in infection of any female patients or resulting children.

DETAILED DESCRIPTION:
This study will enroll couples who wish to have a child in which the man is HIV-seropositive and the woman is HIV-seronegative. The couple will be counseled about their reproductive options, including in vitro fertilization (IVF) donor insemination and adoption. The male patient will be using appropriate therapy to reduce the virus in his semen. Semen will undergo specialized washing to reduce viral contamination of sperm. The sperm are first separated from leukocytes and other seminal constituents by centrifugation over a stepwise gradient. Motile sperm will be separated from the resulting pellet by a swim-up step in which washed sperm are overlaid with fresh medium into which sperm migrate. The final sperm suspension will be stored while testing for HIV is performed by reverse transcription polymerase chain reaction (RT-PCR). Specimens found negative for HIV will then be used for IUI (review: Gilling-Smith et al, 2006; Bujan et al 2007). There is presumably some risk of HIV transmission to the woman and resulting child with this approach; however, over 4000 inseminations reported in Europe over the last 15 years have not resulted in infection of any female patient or resulting child. The woman will be followed for a year after the final IUI to assess seroconversion. If a child is born, he or she will be tested for HIV at 3 months of age.

ELIGIBILITY:
Inclusion Criteria:

Couple must:

* attest to safe sex practices
* know the HIV-status of their partner
* be informed of risks of this procedure and alternatives, including donor insemination
* have the ability to provide informed consent
* been referred or self-refer to Dr. Schust for infertility treatment

Female must:

* be 18-38 years of age
* have a normal menstrual cycle before the IUI cycle
* be negative for HIV, gonorrhea, chlamydia, syphilis, hepatitis B and hepatitis C
* have a standard infertility evaluation and be a candidate for intrauterine insemination

Male must:

* be at least 18 years of age
* be HIV-seropositive
* be under the care of an infectious disease specialist
* disease must be under control without evidence of acquired immunodeficiency syndrome (AIDS), with viral load <50,000 copies/mL and CD4 count > 250 cells/mL for the preceding 6 month period
* have semen quality adequate for intrauterine insemination

If the couple does not achieve pregnancy after IUI, they may continue in the study for 5 additional treatment subsequent cycles. The man must continue to receive care for his HIV and the disease must continue to be under control. Before each cycle of insemination, the couple must each sign an attestation statement that he/she is following safe sex practices, and have repeat testing for sexually-transmitted infections.

Ages: 18 Years to 38 Years | Sex: All
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Danny J Schust, MD, Principal Investigator — University of Missouri-Columbia; Erma Z Drobnis, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Missouri Center for Reproductive Medicine & Fertility, Columbia, Missouri, United States

REFERENCES:
- [Background] Bujan L, Pasquier C, Labeyrie E, Lanusse-Crousse P, Morucci M, Daudin M. Insemination with isolated and virologically tested spermatozoa is a safe way for human immunodeficiency type 1 virus-serodiscordant couples with an infected male partner to have a child. Fertil Steril. 2004 Oct;82(4):857-62. doi: 10.1016/j.fertnstert.2004.02.128. PMID 15482760
- [Background] Bujan L, Hollander L, Coudert M, Gilling-Smith C, Vucetich A, Guibert J, Vernazza P, Ohl J, Weigel M, Englert Y, Semprini AE; CREAThE network. Safety and efficacy of sperm washing in HIV-1-serodiscordant couples where the male is infected: results from the European CREAThE network. AIDS. 2007 Sep 12;21(14):1909-14. doi: 10.1097/QAD.0b013e3282703879. PMID 17721098
- [Background] Chen JL, Philips KA, Kanouse DE, Collins RL, Miu A. Fertility desires and intentions of HIV-positive men and women. Fam Plann Perspect. 2001 Jul-Aug;33(4):144-52, 165. PMID 11496931
- [Background] Gilling-Smith C, Nicopoullos JD, Semprini AE, Frodsham LC. HIV and reproductive care--a review of current practice. BJOG. 2006 Aug;113(8):869-78. doi: 10.1111/j.1471-0528.2006.00960.x. Epub 2006 Jun 2. PMID 16753050
- [Background] Gilling-Smith C, Smith JR, Semprini AE. HIV and infertility: time to treat. There's no justification for denying treatment to parents who are HIV positive. BMJ. 2001 Mar 10;322(7286):566-7. doi: 10.1136/bmj.322.7286.566. No abstract available. PMID 11238138
- [Background] Englert Y, Van Vooren JP, Place I, Liesnard C, Laruelle C, Delbaere A. ART in HIV-infected couples: has the time come for a change of attitude? Hum Reprod. 2001 Jul;16(7):1309-15. doi: 10.1093/humrep/16.7.1309. PMID 11425804
- [Background] Ethics Committee of the American Society for Reproductive Medicine. Human immunodeficiency virus and infertility treatment. Fertil Steril. 2002 Feb;77(2):218-22. doi: 10.1016/s0015-0282(01)03000-x. No abstract available. PMID 11821074
- [Background] Kim LU, Johnson MR, Barton S, Nelson MR, Sontag G, Smith JR, Gotch FM, Gilmour JW. Evaluation of sperm washing as a potential method of reducing HIV transmission in HIV-discordant couples wishing to have children. AIDS. 1999 Apr 16;13(6):645-51. doi: 10.1097/00002030-199904160-00004. PMID 10397558
- [Background] Leruez-Ville M, de Almeida M, Tachet A, Dulioust E, Guibert J, Mandelbrot L, Salmon D, Jouannet P, Rouzioux C. Assisted reproduction in HIV-1-serodifferent couples: the need for viral validation of processed semen. AIDS. 2002 Nov 22;16(17):2267-73. doi: 10.1097/00002030-200211220-00006. PMID 12441798
- [Background] Lesage B, Vannin AS, Emiliani S, Debaisieux L, Englert Y, Liesnard C. Development and evaluation of a qualitative reverse-transcriptase nested polymerase chain reaction protocol for same-day viral validation of human immunodeficiency virus type 1 ribonucleic acid in processed semen. Fertil Steril. 2006 Jul;86(1):121-8. doi: 10.1016/j.fertnstert.2005.12.021. Epub 2006 Jun 6. PMID 16756977
- [Background] Marina S, Marina F, Alcolea R, Exposito R, Huguet J, Nadal J, Verges A. Human immunodeficiency virus type 1--serodiscordant couples can bear healthy children after undergoing intrauterine insemination. Fertil Steril. 1998 Jul;70(1):35-9. doi: 10.1016/s0015-0282(98)00102-2. PMID 9660417
- [Background] Mandelbrot L, Heard I, Henrion-Geant E, Henrion R. Natural conception in HIV-negative women with HIV-infected partners. Lancet. 1997 Mar 22;349(9055):850-1. doi: 10.1016/S0140-6736(05)61754-0. No abstract available. PMID 9121267
- [Background] Pasquier C, Anderson D, Andreutti-Zaugg C, Baume-Berkenbosch R, Damond F, Devaux A, Englert Y, Galimand J, Gilling-Smith C, Guist'hau O, Hollander L, Leruez-Ville M, Lesage B, Maillard A, Marcelin AG, Schmitt MP, Semprini A, Vourliotis M, Xu C, Bujan L; CREAThE Network. Multicenter quality control of the detection of HIV-1 genome in semen before medically assisted procreation. J Med Virol. 2006 Jul;78(7):877-82. doi: 10.1002/jmv.20636. PMID 16721844
- [Background] Politch JA, Mayer KH, Anderson DJ. Depletion of CD4+ T cells in semen during HIV infection and their restoration following antiretroviral therapy. J Acquir Immune Defic Syndr. 2009 Mar 1;50(3):283-9. doi: 10.1097/QAI.0b013e3181989870. PMID 19194315
- [Background] Politch JA, Xu C, Tucker L, Anderson DJ. Separation of human immunodeficiency virus type 1 from motile sperm by the double tube gradient method versus other methods. Fertil Steril. 2004 Feb;81(2):440-7. doi: 10.1016/j.fertnstert.2003.06.028. PMID 14967387
- [Background] Quayle AJ, Xu C, Tucker L, Anderson DJ. The case against an association between HIV-1 and sperm: molecular evidence. J Reprod Immunol. 1998 Dec;41(1-2):127-36. doi: 10.1016/s0165-0378(98)00053-9. PMID 10213305
- [Background] Quayle AJ, Xu C, Mayer KH, Anderson DJ. T lymphocytes and macrophages, but not motile spermatozoa, are a significant source of human immunodeficiency virus in semen. J Infect Dis. 1997 Oct;176(4):960-8. doi: 10.1086/516541. PMID 9333154
- [Background] Sauer MV. Sperm washing techniques address the fertility needs of HIV-seropositive men: a clinical review. Reprod Biomed Online. 2005 Jan;10(1):135-40. doi: 10.1016/s1472-6483(10)60815-2. PMID 15705311
- [Background] Semprini AE, Levi-Setti P, Bozzo M, Ravizza M, Taglioretti A, Sulpizio P, Albani E, Oneta M, Pardi G. Insemination of HIV-negative women with processed semen of HIV-positive partners. Lancet. 1992 Nov 28;340(8831):1317-9. doi: 10.1016/0140-6736(92)92495-2. PMID 1360037
- [Background] Semprini AE, Bujan L, Englert Y, Smith CG, Guibert J, Hollander L, Ohl J, Vernazza P. Establishing the safety profile of sperm washing followed by ART for the treatment of HIV discordant couples wishing to conceive. Hum Reprod. 2007 Oct;22(10):2793-4; author reply 2794-5. doi: 10.1093/humrep/dem197. Epub 2007 Jul 3. No abstract available. PMID 17609245
- [Background] Smith JR, Forster GE, Kitchen VS, Hooi YS, Munday PE, Paintin DB. Infertility management in HIV positive couples: a dilemma. BMJ. 1991 Jun 15;302(6790):1447-50. doi: 10.1136/bmj.302.6790.1447. No abstract available. PMID 2070114
- [Background] Sunderam S, Hollander L, Macaluso M, Vucetich A, Jamieson DJ, Osimo F, Duerr A, Semprini AE. Safe conception for HIV discordant couples through sperm-washing: experience and perceptions of patients in Milan, Italy. Reprod Health Matters. 2008 May;16(31):211-9. doi: 10.1016/S0968-8080(08)31342-1. PMID 18513622
- [Background] Vernazza PL, Gilliam BL, Dyer J, Fiscus SA, Eron JJ, Frank AC, Cohen MS. Quantification of HIV in semen: correlation with antiviral treatment and immune status. AIDS. 1997 Jul;11(8):987-93. PMID 9223732
- [Background] Centers for Disease Control (CDC). Semen banking, organ and tissue transplantation, and HIV antibody testing. MMWR Morb Mortal Wkly Rep. 1988 Feb 5;37(4):57-8, 63. No abstract available. PMID 3122014
- [Background] Centers for Disease Control (CDC). HIV-1 infection and artificial insemination with processed semen. MMWR Morb Mortal Wkly Rep. 1990 Apr 20;39(15):249, 255-6. No abstract available. PMID 2109169
- [Background] Centers for Disease Control and Prevention. Revised guidelines for HIV counseling, testing, and referral. MMWR Recomm Rep. 2001 Nov 9;50(RR-19):1-57; quiz CE1-19a1-CE6-19a1. PMID 11718472